CLINICAL TRIAL: NCT07002203
Title: A Phase Ib Clinical Study of Personalized Neoantigen Peptide Vaccines for Solid Tumors
Brief Title: Personalized Neoantigen Peptide Vaccines for Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seqker Biosciences, Inc. (Industry)
Collaborators: Bumrungrad International Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SQK01-002
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors; Advanced Cancer; Recurrent Cancer; Neoantigen-Specific Immunotherapy; Personalized Cancer Vaccine
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized Neoantigen Peptide Vaccine + Poly-ICLC + Anti-PD-1 (Experimental)
  Interventions: Biological: Personalized Neoantigen Peptide Vaccine

INTERVENTIONS:
Biological: Personalized Neoantigen Peptide Vaccine — This is a personalized cancer vaccine made of 10-20 synthetic long peptides derived from the unique mutations (neoantigens) found in a patient's tumor. Each vaccine is custom-formulated based on whole exome and RNA sequencing of tumor and normal tissue. The peptides are administered intramuscularly in combination with poly-ICLC (Hiltonol) as an adjuvant to enhance immune response. The intervention aims to induce T-cell responses against tumor-specific neoantigens. Vaccinations are given during priming and booster phases, with long-term follow-up and immune monitoring.

SUMMARY:
This clinical trial is studying the safety and efficacy of a personalized cancer vaccine called a neoantigen peptide vaccine in patients with solid tumors. These vaccines are custom-made for each patient using specific mutations (neoantigens) found in their own tumor. The goal is to help the patient's immune system recognize and attack their cancer.

The study will enroll adult patients (20 years or older) who have solid tumors that meet specific stage-related criteria. These include advanced cancers that are resistant to prior treatments and early-stage cancers at high risk of recurrence, where there are no standard adjuvant therapies available.

Participants will receive:

* A personalized neoantigen peptide vaccine designed from the mutations in their tumor tissue.
* Poly-ICLC (Hiltonol), a substance that stimulates the immune system.
* An anti-PD-1 immune checkpoint inhibitor, a drug that helps the immune system stay active against cancer.

The vaccine and drugs will be given through multiple injections over several months. Blood samples and imaging will be used to monitor the immune response and how the cancer responds to treatment. Participants will be followed for up to 12 months.

This study does not include a placebo group. Every participant will receive the personalized vaccine along with the other therapies.

The primary objectives of this study are:

1. To assess whether the treatment is safe and tolerable.
2. To evaluate whether this approach helps control the cancer and can be combined with other standard treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 years or older.
2. Language proficiency: Able to read and understand Thai clearly.
3. Consent: Willing to provide informed consent and sign a participation agreement.
4. Life expectancy: Estimated to be at least 6 months from the date of consent.
5. Eligibility from prior research: Must have participated in the SQK01-002A research project and have tumor tissue confirmed as suitable for neoantigen peptide vaccine production.
6. Performance status: ECOG performance status of 0-2 with stable organ function, no rapid disease progression, or impending organ failure.
7. Cancer diagnosis: Clinically and pathologically confirmed cancer diagnosis, with supporting radiological evidence.
8. Cancer stage-specific criteria:

   i. Advanced cancer: Suitable for immune checkpoint inhibitors (ICIs) and shows resistance to prior therapies, with measurable lesions based on mRECIST1.1 criteria.

   ii. Early-stage cancer: High recurrence risk despite prior surgery and/or radiotherapy, with no current adjuvant treatment standard.
9. Laboratory parameters:

   i. Lymphocyte count ≥ 800 cells/μL. ii. Neutrophil count ≥ 1,500 cells/μL. iii. Platelet count ≥ 75,000 cells/μL. iv. AST ≤ 2.5 times the upper limit of normal (ULN). v. ALT ≤ 2.5 times ULN. vi. Total bilirubin ≤ 1.5 times ULN. vii. Serum creatinine ≤ 1.5 times ULN.
10. Consent to Avoid Pregnancy or Causing Pregnancy Under the Following Criteria i. Female participants not of reproductive age, defined as having undergone a hysterectomy and/or bilateral oophorectomy, experiencing continuous menopause for more than 12 months, or being over 60 years of age.

ii. Female participants of reproductive age must undergo a pregnancy test and have a confirmed negative result during the preparation phase and before the first day of vaccination. They must also consent to using contraception with an efficacy rate greater than 99%, as recommended by the principal investigator, throughout the study duration, including the preparation phase and follow-up, and up to 120 days after the final treatment.

iii. Male participants must consent to using contraception with an efficacy rate greater than 99%, as recommended by the principal investigator, throughout the study duration, including the preparation phase and up to 120 days after the final treatment.

Exclusion Criteria:

1. History of hypersensitivity to peptide vaccines or related substances.
2. Autoimmune disease history.
3. Previous treatments that significantly suppress or impair immune function.
4. Refusal of current standard-of-care treatment.
5. Active brain or central nervous system metastases unless well-controlled with steroids ≤ 10 mg/day prednisolone.
6. Presence of more than one active cancer type.
7. Uncontrolled cardiac conditions, such as unstable angina or advanced heart failure (NYHA Class III/IV).

   i. Participants with pacemakers may be eligible if stabilized for at least 1 month before vaccination.
8. Receipt of any other vaccines within 28 days before the first neoantigen peptide vaccine.
9. Participation in another clinical trial.
10. Use of immunosuppressive drugs or steroids > 10 mg/day prednisolone (except inhaled/intranasal corticosteroids).
11. Pre-existing conditions that could compromise the efficacy or safety of the peptide vaccine.
12. Pregnancy or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | From first vaccination through 72 weeks
  Number and severity of treatment-emergent adverse events, graded according to CTCAE v5.0, to evaluate the safety and tolerability of personalized neoantigen peptide vaccines in combination with poly-ICLC and an anti-PD-1 immune checkpoint inhibitor.

SECONDARY OUTCOMES:
Objective Tumor Response Rate (ORR) | Baseline to 72 weeks after initial vaccination
  Proportion of participants achieving complete or partial response as assessed by RECIST v1.1 or mRECIST criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Horizon Cancer Excellence Center, Bumrungrad International Hospital, Bangkok
  - Phyathai-1 Hospital, Bangkok